CLINICAL TRIAL: NCT04929717
Title: The Effect of Social Media Based Support on Breastfeeding Self-efficacy of Women: A Randomized Controlled Trial
Brief Title: Social Media and Breastfeeding Self Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/06-15
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Breastfeeding
Keywords: breastfeeding self-efficacy; breastfeeding support; social media; WhatsApp
MeSH Terms: conditions — Breast Feeding | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The personal information form and BSES-SF were administered to women in the hospital before the intervention. Breastfeeding education and counseling were provided via social media (WhatsApp) to support women for breastfeeding and to ensure the continuity of breastfeeding in the postpartum period. Breastfeeding education was given to women in the first four weeks after discharge from the hospital. After the breastfeeding education was completed via social media, the counseling process started. Counseling was conducted via social media with a question-answer method between the first and 6th months of postpartum.
  Interventions: Other: Breastfeeding education and counseling; Other: Routine postpartum breastfeeding training included in the hospital procedure
- Control (Other): The women in the control group were pre-tested at the hospital before discharge. The BSES-SF was re-administered by phone at the 3rd and 6th postpartum months. The control group received the routine breastfeeding postpartum educational training given to all women by healthcare personnel as part of the hospital procedures. Except for routine breastfeeding training, no intervention was applied to the control group.
  Interventions: Other: Routine postpartum breastfeeding training included in the hospital procedure

INTERVENTIONS:
Other: Breastfeeding education and counseling — Breastfeeding education was applied for four weeks.
  Arms: Intervention
Other: Routine postpartum breastfeeding training included in the hospital procedure — The routine breastfeeding postpartum educational training given to all women by healthcare personnel as part of the hospital procedures.

SUMMARY:
This study aimed to determine the effect of breastfeeding support on women's breastfeeding self-efficacy via social media. This study was conducted maternity unit at a state hospital in Turkey. Education and consulting about breastfeeding were given via WhatsApp application to women in the intervention group. Women in the control group receive only routine breastfeeding training.

DETAILED DESCRIPTION:
The research was conducted as a randomized controlled trial. The stratified and permutation block randomization methods were used in the study. The personal information form and BSES-SF were administered to women in the hospital before the intervention. Breastfeeding education and counseling were provided via social media (WhatsApp) to support women for breastfeeding and to ensure the continuity of breastfeeding in the postpartum period. Breastfeeding education was given to women in the first four weeks after discharge from the hospital. The control group received the routine breastfeeding postpartum educational training given to all women by healthcare personnel as part of the hospital procedures. Except for routine breastfeeding training, no intervention was applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* being primipara
* being 18 years of age or older
* using the WhatsApp social media application
* having a newborn with a weight of 2500 grams and above
* agreeing to participate in the study

Exclusion Criteria:

* being multiparity
* having a physical or mental health problem that would prevent breastfeeding
* preterm labor (before 37 weeks)
* difficult labor
* either mother or baby having a health problem after birth
* mother's substance use (drug, smoking or alcohol)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All of the people included in the study are female.
Enrollment: 68 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | Baseline
  The scale consists of 14 questions and is a five-point Likert type. The lowest score of 14 points and the highest of 70 points are obtained from the scale. The higher the score indicates a higher self-efficacy perception.
The Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | 3rd month
  The scale consists of 14 questions and is a five-point Likert type. The lowest score of 14 points and the highest of 70 points are obtained from the scale. The higher the score indicates a higher self-efficacy perception.
The Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | 6th month
  The scale consists of 14 questions and is a five-point Likert type. The lowest score of 14 points and the highest of 70 points are obtained from the scale. The higher the score indicates a higher self-efficacy perception.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Ayaz-Alkaya, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)